CLINICAL TRIAL: NCT06576726
Title: Sensorimotor and Psychosocial Trajectories in Adolescents With Tic Disorder
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David Isaacs, Assistant Professor of Neurology and Pediatrics, Vanderbilt University Medical Center
Other Study IDs: 241465
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Tourette Syndrome; Tic Disorder
Keywords: Tourette syndrome; tic disorder; sensorimotor; sensory; motor; sensory over-responsivity; psychosocial; development; behavioral; neurophysiology
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders; Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- adolescents with tic disorder
  Interventions: Other: This study involves no intervention.
- neurotypical adolescents (controls)
  Interventions: Other: This study involves no intervention.

INTERVENTIONS:
Other: This study involves no intervention. — This study involves no intervention.

SUMMARY:
Individuals with tic disorders have lower quality of life, sensory and movement difficulties, and poorer mental, social, and physical health compared to the general population. Current clinical care for individuals with tic disorders is limited: no interventions are proven to prevent or stop the disorder exist, and most treatments focus solely on tics, though other symptoms often affect quality of life more than tics. To develop new treatments and improve care for people with tics, researchers need to better understand the different symptoms people experience and how the brain causes these symptoms.

Many individuals with tic disorders have sensory and movement symptoms other than tics. A common sensory symptom is increased sensitivity to common sensations, such as glare from sunlight, tags in shirt collars, and noises from passing cars. A common movement symptom is poor handwriting and/or poor coordination. In one study of adolescents with tic disorder, difficulty with hand coordination predicted tic severity 7.5 years later, suggesting that sensory and/or motor difficulties may be a risk factor for more severe tics later in life. Despite how common they are, much is unknown about sensory and motor difficulties experienced by people with tic disorders.

Additionally, most studies of people with tics enroll younger children. As a result, little is known about sensory, motor, and psychosocial development in adolescents with tics. Knowledge of sensory and motor difficulties in adolescents with tics is important to understand because, in other adolescent populations, such difficulties are associated with worse mental and social health and worse quality of life. Deepening insight into the sensory, motor, and psychosocial development of adolescents with tic disorders is crucial to identify causes and risk factors for poor health in this population.

The goals of this study are to measure sensory and motor symptoms and function in adolescents with tics and to compare them to adolescents without tics. The research team will enroll adolescents with tics and adolescents without tics to participate in the study. Adolescent participants will complete questionnaires, electroencephalogram (EEG) tasks, and other sensory and motor tasks at baseline (with 2 study visits occurring within 30 days of each other) and 2 years later (again, with 2 study visits, occurring within 30 days of each other). A parent or other adult who knows the adolescent well will also complete questionnaires as part of the study.

DETAILED DESCRIPTION:
The study consists of 4 visits over the course of 2 years. The first 2 visits will occur within 30 days of each other, and then, two years later, participants will be asked to attend two more study visits (again within 30 days of each other).

Study Visit 1 can occur in-person or remotely. If you and your adolescent prefer the remote visit, this will be conducted over Zoom, Microsoft Teams, or another commercial audiovisual platform. During Visit 1, adolescents will be interviewed by a trained rater to assess for tics, obsessive-compulsive disorder (OCD), and attention-deficit/hyperactivity disorder (ADHD). The interview will take about 1 hour. Adolescents will then be asked to complete a series of online questionnaires, asking about sensory experiences, coordination, puberty, mental health, and social health. The questionnaires will take about 1.5 hours to complete. In total Visit 1 will take about 2 hours and 30 minutes.

Study Visit 2 will occur in-person within 30 days of Visit 1. During Visit 2, adolescents will complete questionnaires about sensory experiences, stress, and other symptoms of tic disorders. Questionnaires will take about 1 hour to complete. Then, adolescents' motor coordination, handwriting, and intelligence will be assessed using various tasks and scales. This will take about 2 hours and 30 minutes. Additionally, adolescents' height, weight, and waste circumference will be measured. At the end of the visit, adolescents who are eligible will have an electroencephalogram (EEG) during which their brain activity will be measured while they experience different sensory stimuli (such as puffs of air, simple sounds) and perform different simple motor tasks (such as tapping). The EEG tasks will take about 1 hour and 30 minutes. In total, Visit 2 will take about 5 hours for adolescents eligible for EEG procedures; Visit 2 will take about 3 hours and 30 minutes for adolescents not eligible for EEG procedures. While the adolescent is being assessed, a parent or other adult caregiver will complete questionnaires about the adolescent and themselves; these questionnaires, which take a total of 2 hours to complete, ask about mental health, social health, and quality of life.

Study Visit 3 will occur 2 years after Study Visit 1. Visit 3 can occur in-person or remotely. Visit 3 procedures are identical to Visit 1 procedures.

Study Visit 4 will occur in-person within 30 days of Visit 3. Visit 4 procedures are identical to Visit 2 procedures.

ELIGIBILITY:
* Inclusion criteria for adolescents with tic disorder:

  * adolescent age 11-17 years of age
  * adolescent diagnosis of chronic tic disorder (Tourette syndrome, chronic motor tic disorder, chronic vocal tic disorder)
  * English-speaking adolescent and caregiver/adult proxy (as validated questionnaires are in English)
  * adolescent and caregiver/adult proxy willingness and ability to complete relevant questionnaires
* Exclusion criteria for for adolescents with tic disorder:

  * cognitive or attentional impairment precluding ability of adolescent or caregiver/adult proxy to complete questionnaires and other study measures
  * adolescent diagnosis of autism spectrum disorder (ASD) or psychotic disorder
  * adolescent diagnosis of pervasive genetic disorder besides chronic tic disorders and their known comorbidities
  * adolescent with severe medical conditions unrelated to chronic tic disorders (e.g. uncontrolled seizures, prominent heart conditions)
  * other variables that might influence ratings outside of the typical presentation of chronic tic disorders
* Additional exclusion criteria for EEG tasks for chronic tic disorder sample**

  * adolescent treatment with stimulant medications or anti-seizure medications within the past 30 days
  * use of marijuana or recreational substances within the past 30 days
  * history of seizure
  * history of hearing loss or abnormalities
  * history of neuropathy or overt sensory deficit
  * history of brain surgery or skull-penetrating/deforming trauma
  * history of stroke, brain cancer, or other significant neurologic illness/disorder ** Individuals excluded based on these criteria are ineligible for the EEG portion of the study but can complete the remainder of the study measures.
* Inclusion criteria for control (neurotypical adolescent) participants

  * adolescent age 11-17 years of age
  * English-speaking adolescent and caregiver/adult proxy (as validated questionnaires are in English)
  * adolescent and caregiver/adult proxy willingness and ability to complete relevant questionnaires
* Exclusion criteria for control sample

  * history of tics, ADHD, OCD, or other significant neurodevelopmental or neuropsychiatric disorder.

    ** Note: adolescents with history of mood or anxiety disorder are eligible.
  * cognitive or attentional impairment precluding ability of adolescent or caregiver/adult proxy to complete questionnaires and other study measures
  * adolescent diagnosis of autism spectrum disorder (ASD) or psychotic disorder
  * adolescent diagnosis of pervasive genetic disorder
  * adolescent with severe medical conditions (e.g. uncontrolled seizures, prominent heart conditions)
  * other variables that might influence ratings
* Additional exclusion criteria for EEG tasks for control sample*

  * adolescent treatment with stimulant medications or anti-seizure medications within the past 30 days
  * use of marijuana or recreational substances within the past 30 days
  * history of seizure
  * history of hearing loss or abnormalities
  * history of neuropathy or overt sensory deficit
  * history of brain surgery or skull-penetrating/deforming trauma
  * history of stroke, brain cancer, or other significant neurologic illness/disorder

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants must be willing to attend Visits 2 and 4 in-person
Sampling Method: Non-Probability Sample
Enrollment: 351 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Adolescent/Adult Sensory Profile (AASP) | from baseline to 2-year follow-up
  validated, 60-item self-report questionnaire assessing sensory experiences
Sensory Perception Quotient | from baseline to 2-year follow-up
  35-item self-report questionnaire assessing self-perceived basic sensory sensitivity
Sensory Gating Inventory | from baseline to 2-year follow-up
  validated, 36-item self-report questionnaire assessing sensory over-responsivity
Adolescent Motor Competence Questionnaire (AMCQ) | from baseline to 2-year follow-up
  validated, 26-item self-report questionnaire assessing self-perceived coordination
Bruininks-Oseretsky Test of Motor Proficiency, 2nd edition (BOT-2) | from baseline to 2-year follow-up
  validated, rater-administered scale assessing motor coordination
Purdue pegboard | from baseline to 2-year follow-up
  validated, rater-administered task assessing manual dexterity and coordination
Vibrotactile battery, with BrainGauge (CM4) | from baseline to 2-year follow-up
  Device- and rater-administered battery assessing several features of vibrotactile threshold perception, including static threshold detection, dynamic threshold detection, amplitude discrimination without and with adaptation, sequential and simultaneous frequency discrimination
Tactile gating indices | from baseline to 2-year follow-up
  Participants will undergo a tactile gating paradigm, while monitored on electroencephalogram (EEG), during which puffs of air will be administered to the index finger.
Contingent negative variation indices | from baseline to 2-year follow-up
  Participants will undergo a contingent negative variation paradigm, while monitored on electroencephalogram (EEG), during which puffs of air will be administered to the index finger, cueing the participant to respond

SECONDARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) | from baseline to 2-year follow-up
  gold-standard semi-structured interview assessing tic severity
Premonitory Urge for Tics Scale (PUTS) | from baseline to 2-year follow-up
  validated, 10-item self-report questionnaire assessing premonitory urge severity
Adult ADHD Self-Report Scale for DSM-V (ASRS-V) | from baseline to 2-year follow-up
  6-item self-report questionnaire assessing ADHD severity
Obsessive-Compulsive Inventory-Child Version-Revised (OCI-CV-R) | from baseline to 2-year follow-up
  validated, 18-item self-report questionnaire assessing OCD symptom severity
PROMIS Pediatric SF GenPop v3.0 - Anxiety 8a | from baseline to 2-year follow-up
  8-item self-report scale assessing anxiety severity
PROMIS Pediatric SF GenPop v3.0 - Depressive Sx 8a | from baseline to 2-year follow-up
  8-item self-report questionnaire assessing depression severity
PROMIS Pediatric SF GenPop v3.0 - Peer Relationships 8a | from baseline to 2-year follow-up
  8-item self-report questionnaire assessing self-perceived peer relationship quality
PROMIS Pediatric SF v1.0 - Family Relationships 8a | from baseline to 2-year follow-up
  8-item self-report questionnaire assessing self-perceived family relationship quality
PROMIS Pediatric SF v1.0 - Sleep Disturbance 8a | from baseline to 2-year follow-up
  8-item self-report questionnaire assessing self-perceived sleep quality
PROMIS Pediatric SF v1.0 - Meaning and Purpose 8a | from baseline to 2-year follow-up
  8-item self-report questionnaire assessing meaning and purpose in life
PROMIS Pediatric SF v1.0 - Life Satisfaction 8a | from baseline to 2-year follow-up
  8-item self-report questionnaire assessing degree of satisfaction with life
Lubben Social Network Scale | from baseline to 2-year follow-up
  12-item self-report scale assessing extent of individual's social network
UCLA Loneliness Scale | from baseline to 2-year follow-up
  20-item self-report scale assessing loneliness
Height, weight, waist measurement | from baseline to 2-year follow-up
  Height, weight, waist measurement
Beery Visuomotor Integration, 6th edition | from baseline to 2-year follow-up
  validated, rater-administered measure assessing visuo-motor integration
Writing kinematic indices | from baseline to 2-year follow-up
  Using MovAlyzeR software program on a Wacom tablet, the participant will perform several writing exercises to quantify writing kinematic characteristics.
Adolescent Stress and Adversity Inventory (STRAIN) | from baseline to 2-year follow-up
  Per the scale developer's website: "The Stress and Adversity Inventory (STRAIN) is an NIMH/RDoC-recommended instrument for efficiently and reliably assessing exposure to acute and chronic life stress over the life course. The measure is entirely online and systematically inquires about a diverse array of acute life events (e.g., deaths of relatives, job losses, negative health events) and chronic difficulties (e.g., ongoing health problems, work problems, relationship problems, financial problems, etc.) that have implications for human health and well-being. Stressors occurring in early life (e.g., childhood maltreatment or neglect, parental loss/separation, etc.) are also queried. Participants are asked to rate the severity, frequency, timing, and duration of each stressor they endorse...Based on this information, the system produces 455 variables that are used to assess an individual's cumulative exposure to stress."
Finger tapping indices | from baseline to 2-year follow-up
  Participants will perform a finger tapping task, while monitored on electroencephalogram (EEG)
Child Behavior Checklist | from baseline to 2-year follow-up
  validated, 113-item, proxy-report questionnaire assessing psychopathology in children and adolescents
Conners-4 | from baseline to 2-year follow-up
  validated, 117-item, proxy-report questionnaire assessing symptoms of ADHD and commonly co-occurring diagnoses of ADHD in children and adolescents
Toronto Obsessive-Compulsive Scale (TOCS) | from baseline to 2-year follow-up
  validated, 21-item proxy-report questionnaire assessing OCD symptom severity
Social Communication Questionnaire - Lifetime | from basline to 2-year follow-up
  validated, 40-item proxy-report questionnaire assessing lifetime history of communication difficulties/differences and other symptoms suggestive of autism spectrum disorder
BRIEF-2 Parent Form | from baseline to 2-year follow-up
  validated, 63-item proxy-report questionnaire assessing executive dysfunction
PedsQL Family Impact Module, Version 2.0 | from baseline to 2-year follow-up
  validated, 36-item proxy-report questionnaire assessing impact of child's/adolescent's health on family
PROMIS Parent Proxy SF GenPop v3.0 - Anxiety 8a | from baseline to 2-year follow-up
  8-item, proxy-report questionnaire assessing anxiety
PROMIS Parent Proxy SF GenPop v3.0 - Depressive Sx 8a | from baseline to 2-year follow-up
  8-item, proxy-report questionnaire assessing depression
PROMIS Parent Proxy SF GenPop v3.0 - Peer Relationships 7a | from baseline to 2-year follow-up
  7-item, proxy-report questionnaire assessing proxy-perceived peer relationship quality
PROMIS EC Parent-Report SF v1.0 - Social Relationships - Family Relationships 4a | from baseline to 2-year follow-up
  4-item, proxy-report questionnaire assessing proxy-perceived family relationship quality
PROMIS EC Parent-Report SF v1.0 - Sleep Health - Disturbance 4a | from baseline to 2-year follow-up
  4-item, proxy-report questionnaire assessing proxy-perceived sleep disturbances
PROMIS Parent Proxy SF v1.0 - Meaning and Purpose 8a | from baseline to 2-year follow-up
  8-item, proxy-report questionnaire assessing proxy-perceived meaning and purpose in adolescent's life
PROMIS Parent Proxy SF v1.0 - Life Satisfaction 8a | from baseline to 2-year follow-up
  8-item, proxy-report questionnaire assessing adolescent's satisfaction with life
Short Sensory Profile - 2 | from baseline to 2-year follow-up
  validated, 34-item proxy-report questionnaire assessing sensory experiences
Developmental Coordination Disorder Questionnaire | from baseline to 2-year follow-up
  15-item proxy-report questionnaire assessing motor coordination

OTHER OUTCOMES:
Edinburgh Handedness Inventory - Short Version | from baseline to 2-year follow-up
  4-item self-report questionnaire to assess extent of individual's left- or right-handed dominance
Pubertal Development Scale | from baseline to 2-year follow-up
  5-item self-report scale assessing pubertal stage, based on self-reported signs
Weschler Abbreviated Scale of Intelligence, 2nd edition (WASI-II), 2-subtest with Vocabulary and Matrix Reasoning | baseline
  validated, rater-administered measure assessing intelligence
UCLA Loneliness Scale (Adult Proxy) | from baseline to 2-year follow-up
  20-item self-report questionnaire assessing loneliness
PROMIS SF v1.0 - Anxiety 8a (Adult Proxy) | from baseline to 2-year follow-up
  8-item, self-report questionnaire assessing adult proxy's anxiety
PROMIS SF v1.0 - Depression 8a (Adult Proxy) | from baseline to 2-year follow-up
  8-item, self-report questionnaire assessing adult proxy's depression
Perceived Stress Scale (Adult Proxy) | from baseline to 2-year follow-up
  10-item self-report questionnaire assessing adult proxy's self-perceived stress
Interpersonal Support Evaluation List (Adult Proxy) | from baseline to 2-year follow-up
  12-item self-report questionnaire assessing adult proxy's self-perceived social support

CONTACTS AND LOCATIONS:
Overall Officials: David Isaacs, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashvile, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided
As per NIH guidelines, de-identified data will be shared in an established repository (https://sharing.nih.gov/data-management-and-sharing-policy/sharing-scientific-data/repositories-for-sharing-scientific-data) no later than 12 months after the end of any proposed funding period or within 12 months of the last study visit, whichever comes first. The data sharing plan is not yet available in an online format.